CLINICAL TRIAL: NCT05945667
Title: Prospective Study on the Efficacy and Safety of Uronext® in Parallel Groups in Women With Cystitis in the Acute Stage
Brief Title: Efficacy and Safety of Uronext® in Women With Cystitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PharmaLinea Ltd. (Industry)
Collaborators: NPO Petrovax Pharm LLC. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UN-1
Record Dates: First submitted 2023-07-06; First posted 2023-07-14 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Cystitis
MeSH Terms: conditions — Cystitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monural (Active Comparator): 3000 mg of fosfomycin trometamol per sachet
  Interventions: Drug: Monural
- UroNext + Monural (Experimental): 3000 mg of fosfomycin trometamol per sachet 500 mg of Qcran, 2000 mg of D-mannose, 5 mcg of vitamin D3 per sachet
  Interventions: Drug: Monural; Dietary Supplement: UroNext

INTERVENTIONS:
Drug: Monural — 1 sachet, only 1st day of trial
Dietary Supplement: UroNext — 1 sachet per day for the first 7 days, followed by 7 days break Same scheme to be repeated for 3 months
  Arms: UroNext + Monural

SUMMARY:
The study is designed as a prospective parallel open label, two-arm, single center study exploring efficacy and safety of the use of the dietary supplement Uronext in women with cystitis in the acute stage. 120 otherwise healthy women with acute cystitis infection confirmed with the urine bacteriological examinations, aged 18-18 years, will be recruited. The distribution of patients will be done in 1:1 ratio. Control group will receive standard therapy, Monural (fosfomycin trometamol) 3 g, at the first day of the trial. The second group will also receive Monural (fosfomycin trometamol) 3 g, at the first day of the trial as well as Uronext food supplement, 1 time per day for the first 7 days. After the 7 day break, participants in the second group will follow supplementation scheme for the next 3 month.

Primary objective of the study is evaluation of the effectiveness of the dietary supplement Uronext in women with cystitis in the acute stage in the prevention of subsequent exacerbations of recurrent cystitis during 3 months of observation, measured as the number of relapses throughout the study period. Participnats will also fill in urination diary and questionnaires related to pain perception, quality of life and cystitis symptoms. Urine samples will be further examined at the follow up visits.

Safety will be evaluated based on reported adverse events, assessment of vital signs and laboratory evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18 and 80.
* Patients who are able to fill out questionnaires, and wish to take part in the study.
* Cystitis in the acute stage.
* Informed consent to participate in the study.
* The patient's willingness and ability to fulfill the requirements of the protocol throughout the study.
* Consent of the patient and partner with preserved reproductive potential to use adequate methods of contraception (for example, a double barrier method) during the entire period of the study (including the period of follow-up).
* The presence of the gynecologist's conclusion obtained within 6 months before the patient's participation in the study about the absence of concomitant pathologies that can distort the results of the study.
* The presence of the results of bacteriological urine tests obtained within 7-10 days before the patient's participation in the study, pathogens of infections of the lower urinary tract. If the results of urine bacteriological examinations are not available, the results of urine culture tests performed at Visit 1 will be taken into account.

Exclusion Criteria:

* Patients with signs of upper urinary tract infection, such as temperature above 38°C, side/lower back pain, or soreness.
* Burdened allergic history.
* Hypersensitivity to any of the components that make up the investigational drugs.
* Patients with congenital anomalies in the development of genitourinary organs (exstrophy of the bladder, hypospadias, epispadias).
* Patients after undergoing surgical interventions on the organs of the genitourinary system.
* Patients who at the time of inclusion in the study noted: neurogenic dysfunction of the bladder, urinary incontinence, sclerosis of the neck of the bladder, urethral stricture, stone / stones of the bladder, bladder cancer, diverticula of the bladder, as well as other diseases of the genitourinary organs requiring specialized treatment.
* Any malignant neoplasm in the anamnesis.
* Unsatisfactory glycemic control (HbA1c ≥8%) in diabetes mellitus.
* Patients with uncontrolled infection as a result of exposure to human immunodeficiency virus (HIV) and/or active hepatitis.
* Patients with a history of drug or alcohol dependence within the last 5 years.
* Any clinically significant condition due to which, according to the researcher, the patient cannot take part in the study;
* Pregnancy, lactation, pregnancy planning during the study.
* Patients with any other serious or uncontrollable physical or mental condition/disease that the Researcher determines may put the patient at high risk of being removed from the study may disrupt or disprove the results of the study or likely prevent the patient from complying with the requirements of the study or completing the study.
* Participation in another clinical trial less than 6 months before the start of the study.
* Any other conditions that the researcher believes may indicate that the patient is not eligible to participate in the study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Cystitis relapses | 3 months
  Proportion of patients who did not have relapses of the disease at Visit 3

SECONDARY OUTCOMES:
Pain intensity on the 100 mm Visual Analog Scale | 3 days
  The sum of the difference in pain intensity on the 100 mm Visual Analog Scale. 0 indicates that the pain isn't bothering, 100 indicates strongly bothering pain.
Urinary urge severity on the 100 mm Visual Analog Scale | 6, 24, 48, and 72 hours
  Urinary urge severity on a 100-mm visual analog scale after initiation of study therapy. 0 indicates that the urinary urge isn't bothering, 100 indicates strongly bothering urinary urge.
Urinary frequency severity on the 100 mm Visual Analog Scale | 6, 24, 48, and 72 hours
  Urinary frequency severity on a 100-mm scale after initiation of study therapy. 0 indicates that the urinary frequency isn't bothering, 100 indicates strongly bothering urinary frequency.
Recurrence rate | 3 months
  Recurrence rate between Visit 1 and Visit 3
Urination frequency | 3 days
  Urination frequency based on the Urination Diary on Days 1, 2, and 3 of observation.
Average urine volume | 3 days
  Average urine volume based on the Urination Diary on Days 1, 2, and 3 of observation.
Microorganism growth in urine culture | 3 months
  Proportion of patients with no microorganism growth in urine culture at Visit 2 and 3
Acute Cystitis Symptom Score Questionnaire - Typical | 3 months
  Change in the Acute Cystitis Symptom Questionnaire score (ACSS) ) - Typical symptoms Likert scale with 6 items; for each item 0 indicates no issues and 3 sever issues
Acute Cystitis Symptom Score Questionnaire (ACSS) - Differential | 3 months
  Change in the Acute Cystitis Symptom Questionnaire score (ACSS) - Differential symptom score Likert scale with 4 items; for each item 0 indicates no issues and 3 sever issues
Acute Cystitis Symptom Score Questionnaire (ACSS) - QoL | 3 months
  Change in the Acute Cystitis Symptom Score Questionnaire (ACSS) - QoL Likert scale with 4 items; for each item 0 indicates not being affected and 3 being extremely affected
Acute Cystitis Symptom Score Questionnaire (ACSS) - Dynamics | 3 months
  Change in the Acute Cystitis Symptom Score Questionnaire (ACSS) - Dynamics
  1 question; 0 indicates feeling back to normal and 4 indicates feeling worse
Quality of Life Visual Analog Scale | 3 months
  Change is Quality of Life Visual Analog Scale score 0 indicates symptomes are not bothering and 10 indicates extreme impact on quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Urology Clinic of Moscow State University of Medicine and Dentistry, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No